CLINICAL TRIAL: NCT00111150
Title: Study of the Safety and Efficacy of Daily Tenofovir Disoproxil Fumarate for the Prevention of HIV Infection in Heterosexually Active Young Adults in Botswana
Brief Title: Botswana Tenofovir Oral HIV Prophylaxis Trial
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Consenting participants entered tenofovir/emtricitabine oral prophylaxis trial
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Botswana Ministry of Health (Other Government); Gilead Sciences (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CDC-NCHSTP-4321; BOTUSA MB04
Record Dates: First submitted 2005-05-17; First posted 2005-05-18 (Estimated); Last update posted 2007-03-19 (Estimated); Status verified 2007-03

CONDITIONS: HIV Infection
Keywords: HIV incidence; HIV prevention
MeSH Terms: conditions — HIV Infections | interventions — Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Tenofovir Disoproxil Fumarate 300 mg daily

SUMMARY:
This study will test whether taking a pill of tenofovir (an antiretroviral medicine) is safe for sexually-active young adults in Botswana without HIV infection and whether it will reduce their risk of getting an HIV infection.

DETAILED DESCRIPTION:
Twelve hundred healthy, sexually active women and men, 18-29 years old, without HIV infection will be enrolled in Francistown and Gaborone, Botswana. They will be provided with free male and female condoms, repeated individualized risk-reduction counseling, diagnosis and treatment of sexually transmitted diseases, and women will be provided with a choice of effective family planning methods. In addition, volunteers will be randomized to receive either Tenofovir or a placebo pill to take once a day. Volunteers will be seen monthly for at least 12 months to monitor for side effects and toxicities and to test their HIV status. Persons who become HIV infected during the trial will receive ongoing supportive counseling, CD4 and viral load monitoring, education about HIV infection/disease, and access to HIV care including free antiretrovirals when clinically indicated. Volunteer safety will be monitored by a local ethics committee, Centers for Disease Control Institutional Review Board (CDC IRB) and an independent data safety and monitoring board.

ELIGIBILITY:
Inclusion Criteria:

* citizen of Botswana 18-29 years old
* sexually active
* HIV uninfected
* Hepatitis B and C uninfected
* Calculated creatinine clearance >= 60 mL/min
* hemoglobin >= 8 gm/dL
* ALT and AST <= 2x ULN
* total bilirubin <= 1.5 mg/dL
* total serum amylase <= 1.5x ULN
* Serum phosphorus >= 2.2 mg/dL
* willing to use effective contraception
* living within 1 hours travel of study clinic
* pass comprehension test
* willing and able to give informed consent

Exclusion Criteria:

* history of significant renal or bone disease
* any chronic illness requiring ongoing prescription medication
* pregnant or breastfeeding
* planning to move away from site in the next year
* participating in another HIV prevention or vaccine safety trial
* any other clinical condition or prior therapy that, in the opinion of the study physician, would make the volunteer unsuitable for the study or unable to comply with the dosing requirements

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1200
Dates: Start 2005-09; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Adverse drug reactions in the tenofovir and placebo arms
HIV incidence in the tenofovir and placebo arms

SECONDARY OUTCOMES:
Changes in levels of unprotected sex during the trial
Adherence to medication
Antiretroviral (ARV) resistance patterns in seroconverters
Viral set point in seroconverters

CONTACTS AND LOCATIONS:
Overall Officials: Dawn K Smith, MD, MS, MPH, Study Chair — CDC and BOTUSA; Lynn A Paxton, MD, MPH, Study Chair — Centers for Disease Control and Prevention
Locations (2):
- Centers for Disease Control and Prevention, Atlanta, Georgia, United States
- BOTUSA HIV Prevention Research Unit, Francistown and Gaborone, Botswana